CLINICAL TRIAL: NCT03195829
Title: A Computerized Cognitive Stimulation Program in Elderly With Mild Cognitive Impairment: A Feasibility Study
Brief Title: Feasibility Study of a Computerized Cognitive Stimulation
Acronym: PSCogStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leila DJABELKHIR (Other)
Responsible Party: Sponsor-Investigator, Leila DJABELKHIR, Neuropsychologist, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUSAGE
Record Dates: First submitted 2017-06-12; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Mild Cognitive Impairment, So Stated
Keywords: Mild Cognitive Impairment; Computerized Cognitive Stimulation; Cognition; Psychosocial factors
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot study, single blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized cognitive stimulation (Experimental): Computerized Cognitive Stimulation was administered to intervention group (IG).
  Interventions: Behavioral: Computerized Cognitive Stimulation
- Multimedia-based internet activities (Active Comparator): Multimedia-based internet activities was administered to active control group (ACG).
  Interventions: Behavioral: Multimedia-based internet

INTERVENTIONS:
Behavioral: Computerized Cognitive Stimulation — The intervention group performed 12-week, 90-minutes per week of cognitive stimulation in group using a tablet with a commercial software with specific exercises to train the cognitive functioning and promote the relation ties in group-session.The program's difficulty level was adjusted to the MMSE score, and was gradually increased.
  Arms: Computerized cognitive stimulation
Behavioral: Multimedia-based internet — The active control group had access to different Multimedia contents (travel, photos, music, TV program, cooking recipes) using a tablet, 90-minutes per week each week during 3-months. Each group session was centered in a particular topic, participants were able to select different media free available in Internet.
  Arms: Multimedia-based internet activities

SUMMARY:
This non-pharmacological interventional feasibility study evaluate a computerized cognitive stimulation program in elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
Involvement in social and leisure activities has been associated with a decreased risk of dementia in the elderly with Mild Cognitive Impairment (MCI). MCI is a crucial phase to prevent the worsening of cognitive decline in elderly at risk to develop dementia. These last years, the use of computerized training programs to enhance cognitive functioning showed positive and promising results. However, the effects on psychosocial factors still poorly documented in cognitive interventions in MCI. It seems essential to promote these factors involving social ties, group dynamic, the motivation, as factors that can contribute to enhance social life and cognitive functioning.

This feasibility study evaluated a computer-based cognitive stimulation in elderly with MCI and explore the effects on cognitive and psychosocial components.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* Absence of history of alcohol or other substance consumption
* No engagement in other cognitive intervention program

Exclusion Criteria:

* Psychiatric and neurological disorders
* Conversion toward dementia during intervention
* Sensory and or motor deficit that could interfere with the use of computer tool

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
GROBER-BUSCHKE TEST | Baseline assessment before intervention, change from baseline at 3 months immediately after intervention
  Assessment of free and cued recall of episodic memory

SECONDARY OUTCOMES:
Technologies Acceptation Questionnaire | Baseline assessment before intervention, change from baseline at 3 months immediately after intervention
  Assessment of acceptability of communication and information technologies

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie AR RIGAUD, Professor, Principal Investigator — Broca University Hospital

IPD SHARING:
Plan to Share IPD: No